CLINICAL TRIAL: NCT01077921
Title: Phase II Study of Propranolol as Anti-Adhesive Therapy for Sickle Cell Disease
Brief Title: Study of Propranolol as Anti-Adhesive Therapy in Sickle Cell Disease (SCD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laura M. De Castro, MD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Laura M. De Castro, MD, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00018427; K01HL096434-02 (NIH); 5R21HL096123-02 (NIH)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Results first posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Sickle Cell Disease
Keywords: sickle; adhesion; propranolol
MeSH Terms: conditions — Anemia, Sickle Cell; Tissue Adhesions | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol (Experimental): Drug arm
  Interventions: Drug: Propranolol
- Sugar pill (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Treatment will be with a standard propranolol dose of 40 mg every 12 hrs.Each patient will participate in 6 weeks of treatment with placebo or study drug (propranolol), followed by a 2-week wash-out period and then 6 weeks of treatment with the other modality (placebo or propranolol).
  Arms: Propranolol
Drug: Placebo — Treatment will be with a standard propranolol dose of 40 mg every 12 hrs.Each patient will participate in 6 weeks of treatment with placebo or study drug (propranolol), followed by a 2-week wash-out period and then 6 weeks of treatment with the other modality (placebo or propranolol).
  Arms: Sugar pill

SUMMARY:
An open label, prospective, randomized cross-over phase II study in up to 60 sickle cell patients who are either homozygous for Hb S or have HbSB0 thalassemia. Initially, each patient will be treated for 6 weeks with placebo or a standard dose of propranolol (40 mg) every 12 hrs. This will be followed by a 2-week washout period after which, patients will receive the other treatment modality (placebo or propranolol).

We Hypothesize that propranolol administered in vivo on a daily basis for 6 weeks (1) will decrease baseline adhesion to endothelial cells and will substantially abrogate epinephrine-stimulated adhesion to endothelial cells, as measured in vitro; (2) will improve biomarkers of endothelial activation and dysfunction; and (3) can be safely used in patients with SCD. Thus, the use of propranolol in SCD may represent a safe and effective means of anti-adhesive therapy in SCD.

Study Objectives:

Primary Objective:

• To establish the safety and efficacy of long-term therapy with propranolol as an anti-adhesive therapy for SCD.

Secondary Objective:

• To evaluate changes in soluble markers of endothelial activation and dysfunction.

Correlative Science Objective:

• To determine whether response to propranolol therapy is associated with polymorphisms in genes encoding the proteins involved in the upregulation of Sickle Red Blood Cell (SS RBC) adhesion by epinephrine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis by electrophoresis (HEP) of Hemoglobin (Hgb) SS or Hgb Sβ0 thalassemia (all patients followed at our clinic have HEP-confirmed diagnosis on file)
* Age ≥ 18 years
* Blood pressure (BP) Systolic ≥ 95mm Hg and Diastolic ≥ 50mm Hg
* Heart rate (HR) ≥ 70 and ≤ 110 bpm
* Oxygen saturation by pulse oximeter and at room air ≥ 92%
* Hematocrit (Hct) ≥ 20% and Hb > 6.0 g/dL
* Euthyroid status as indicated by normal Thyroid Stimulating Hormone (TSH)
* SS RBCs obtained during screening period demonstrating an adhesion response to epinephrine of 40% over non-stimulated baseline adhesion to endothelial cells
* Capacity to understand and sign informed consent

Exclusion Criteria:

* History of vaso-occlusive episode during the 6 wks prior to screening
* RBC transfusion during the 3 months prior to study entry
* Ongoing pregnancy
* History of heart failure, myocardial infarct (MI), bradyarrhythmias, conduction defects
* History of asthma or reactive airway disease
* History of thyroid disease
* Diabetes
* Renal insufficiency (BUN >21 mg/dL and/or Creatinine >1.4 mg/dL)
* Use during the screening or study period of any of the following medications: antihypertensives, diuretics, thyroid replacement therapy, anti-arrhythmia medications, bronchodilators, inhaled steroids, insulin, or hypoglycemic medication
* History of allergy to sulfonamides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Zennadi R, Hines PC, De Castro LM, Cartron JP, Parise LV, Telen MJ. Epinephrine acts through erythroid signaling pathways to activate sickle cell adhesion to endothelium via LW-alphavbeta3 interactions. Blood. 2004 Dec 1;104(12):3774-81. doi: 10.1182/blood-2004-01-0042. Epub 2004 Aug 12. PMID 15308566
- [Background] Zennadi R, Moeller BJ, Whalen EJ, Batchvarova M, Xu K, Shan S, Delahunty M, Dewhirst MW, Telen MJ. Epinephrine-induced activation of LW-mediated sickle cell adhesion and vaso-occlusion in vivo. Blood. 2007 Oct 1;110(7):2708-17. doi: 10.1182/blood-2006-11-056101. Epub 2007 Jul 3. PMID 17609430
- [Background] Zennadi R, Chien A, Xu K, Batchvarova M, Telen MJ. Sickle red cells induce adhesion of lymphocytes and monocytes to endothelium. Blood. 2008 Oct 15;112(8):3474-83. doi: 10.1182/blood-2008-01-134346. Epub 2008 Jul 29. PMID 18664622
- [Background] Eyler CE, Jackson T, Elliott LE, De Castro LM, Jonassaint J, Ashley-Koch A, Telen MJ. beta(2)-Adrenergic receptor and adenylate cyclase gene polymorphisms affect sickle red cell adhesion. Br J Haematol. 2008 Apr;141(1):105-8. doi: 10.1111/j.1365-2141.2008.07008.x. PMID 18324973
- [Background] De Castro LM, Zennadi R, Jonassaint JC, Batchvarova M, Telen MJ. Effect of propranolol as antiadhesive therapy in sickle cell disease. Clin Transl Sci. 2012 Dec;5(6):437-44. doi: 10.1111/cts.12005. Epub 2012 Oct 17. PMID 23253664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Duke adult sickle cell clinic. Those that consented underwent a screening visit to determine eligibility. If eligible they were enrolled on the study and received study drug within 30 days of screening
Pre-assignment Details: Eighty-four patients were approached for the study, of those 28 declined to participate, 14 remained undecided. Forty-two patients consented. Thirthy-one of those consenting were enrolled and 27 randomized to the study.
Groups:
- Propranolol-first: Cross-over study comprising treatment with propranolol for 6 weeks with a standard dose of 40 mg every 12 hrs, followed by a 2 weeks period washout, then similar treatment period with placebo followed by another 2 weeks washout period
- Placebo-first: Cross-over study comprising treatment with placebo for 6 weeks, followed by a 2 weeks period washout, then similar treatment period with propranolol with a standard dose of 40 mg every 12 hrs., followed by another 2 weeks washout period.
Period: First Intervention
Arm/Group | Propranolol-first | Placebo-first
Started | 14 | 13
Completed | 13 | 12
Not Completed | 1 | 1
Period: Washout
Arm/Group | Propranolol-first | Placebo-first
Started | 13 | 12
Completed | 13 | 10
Not Completed | 0 | 2
Period: Second Intervention
Arm/Group | Propranolol-first | Placebo-first
Started | 13 | 10
Completed | 13 | 9
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol-first | Placebo-first | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.2 [29.4 to 40.8] | 26.1 [24.7 to 32.7] | 30.4 [25.6 to 39.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: SS RBC Adhesion (Epi -1d/cm2- vs. Sham) by Treatment
Description: The stickiness of SS RBC will be evaluated by a well-established in vitro assay of adhesion of SS RBCs to cultured endothelial cells using a flow chamber. Overall change of adhesion from baseline to post intervention( Week 0 to 6 and week 8 to 14) in unstimulated cells (Sham treated) vs. Stimulated Red Blood Cells (Epi-treated) at 1 dyne/cm2
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Mean (Standard Deviation); unit: Percentage of total RBC
Groups:
- Propranolol: All subjects completing the propranolol treatment phase.
- Placebo: All subjects completing the placebo treatment phase.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
Percentage of total RBC
  Epinephrine Treated Red blood cells | 0 (24.4) | -0.3 (20.1)
  unstimulated cells (Sham treated) | 7.4 (18.7) | 2.7 (26)

2. Secondary Outcome: Overall Change of Plasma Levels of sE-selectin
Description: Biomarkers of Endothelial Activation and Dysfunction: Overall change of Plasma levels of sE-selectin measured in triplicate on plasma samples using commercially available ELISA kits from baseline to post intervention ( Week 0 to 6 and week 8 to 14).
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Placebo: All subjects completing placebo treatment phase.
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
ng/ml | -3.9 (12.1) | 3.7 (9.3)

3. Primary Outcome: SS RBC Adhesion (Epi -2d/cm2- vs. Sham) by Treatment
Description: The stickiness of SS RBC will be evaluated by a well-established in vitro assay of adhesion of SS RBCs to cultured endothelial cells using a flow chamber. Overall change of adhesion from baseline to post intervention( Week 0 to 6 and week 8 to 14) in unstimulated cells (Sham treated) vs. Stimulated Red Blood Cells (Epi-treated) at 2 dyne/cm2
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Mean (Standard Deviation); unit: Percentage of total RBC
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
Percentage of total RBC
  Epi-treated Red blood cells | 0.2 (13.8) | -2.8 (10.7)
  unstimulated cells (Sham treated) | 2.7 (11.2) | 4.4 (13)

4. Primary Outcome: SS RBC Adhesion (Epi -3d/cm2- vs. Sham) by Treatment
Description: The stickiness of SS RBC will be evaluated by a well-established in vitro assay of adhesion of SS RBCs to cultured endothelial cells using a flow chamber. Overall change of adhesion from baseline to post intervention( Week 0 to 6 and week 8 to 14) in unstimulated cells (Sham treated) vs. Stimulated Red Blood Cells (Epi-treated) at 3 dyne/cm2
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Mean (Standard Deviation); unit: Percentage of total RBC
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
Percentage of total RBC
  Epi-treated Red blood cells | 0.5 (9.7) | -2.8 (7.5)
  unstimulated cells (Sham treated) | -0.1 (9.3) | 4.3 (10)

5. Secondary Outcome: Overall Change of Plasma Levels of sP-selectin
Description: Biomarkers of Endothelial Activation and Dysfunction: Overall change of Plasma levels of sP-selectin measured in triplicate on plasma samples using commercially available ELISA kits from baseline to post intervention ( Week 0 to 6 and weeks 8 to 14).
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
ng/ml | -5 (13.9) | -12.8 (54.8)

6. Secondary Outcome: Overall Change of Plasma Levels of sICAM-1
Description: Biomarkers of Endothelial Activation and Dysfunction: Overall change of Plasma levels of sICAM-1 measured in triplicate on plasma samples using commercially available ELISA kits from baseline to post intervention ( Week 0 to 6 and week 8 to 14)
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
ng/ml | -6.4 (15.3) | 5.4 (28.5)

7. Secondary Outcome: Overall Change of Plasma Levels of sVCAM-1
Description: Biomarkers of Endothelial Activation and Dysfunction: Overall change of Plasma levels of sVCAM-1 measured in triplicate on plasma samples using commercially available ELISA kits from baseline to post intervention ( Week 0 to 6 or week 8 to 14)
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
ng/ml | -16.7 (144.2) | -7.2 (117.7)

8. Secondary Outcome: Overall Change of Hemoglobin (Hgb) Levels
Description: Overall change of Hemoglobin (Hgb) levels from baseline to post intervention( Week 0 to 6 and week 8 to 14) Placebo vs. Propranolol treated
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Median (Inter-Quartile Range); unit: gm/dL
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
gm/dL | 0.2 [0.1 to 0.5] | -0.1 [-0.7 to 0.4]

9. Secondary Outcome: Overall Change of Hematocrit (Hct) Levels
Description: Overall change of Hematocrit (Hct) levels from baseline to post intervention( Week 0 to 6 and week 8 to 14) Placebo vs. Propranolol treated
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Median (Inter-Quartile Range); unit: percentage of red blood cells
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
percentage of red blood cells | 1 [0 to 2.0] | 0 [-2.0 to 1.0]

10. Secondary Outcome: Overall Change of Lactate Dehydrogenase (LDH) Levels
Description: Overall change of LDH levels from baseline to post intervention( Week 0 to 6 and week 8 to 14) Placebo vs. Propranolol treated
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
IU/L | 24 [-69 to 107] | -5 [-40.5 to 33]

11. Secondary Outcome: Overall Change of Oxygen Saturation (02Sat) Levels
Description: Overall change of Oxygen Saturation (02Sat) levels from baseline to post intervention( Week 0 to 6 and week 8 to 14) Placebo vs. Propranolol treated
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Median (Inter-Quartile Range); unit: percentage of oxygen saturation
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
percentage of oxygen saturation | 0 [0 to 2] | 0 [-1 to 1.5]

12. Secondary Outcome: Overall Change of Systolic Blood Pressure Levels
Description: Overall change of Systolic Blood Pressure levels from baseline to post intervention (Week 0 to 6 and week 8 to 14) Placebo vs. Propranolol treated
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
mmHg | -1.0 [-4.0 to 5.0] | -1.0 [-8.0 to 5.5]

13. Secondary Outcome: Overall Change of Diastolic Blood Pressure Levels
Description: Overall change of Diastolic Blood Pressure levels from baseline to post intervention (Week 0 to 6 and week 8 to 14) Placebo vs. Propranolol treated
Time Frame: Week 0 to 6 and week 8 to 14
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 22 | 23
mmHg | 0 [-4.0 to 5.0] | -1 [-7.0 to 5.0]

ADVERSE EVENTS:
Description: All patients who were enrolled and had at least one baseline visit are included in the "at risk" category.
Arm/Group | Propranolol | Placebo
Serious Adverse Events (participants affected / at risk) | 4/27 | 3/27
Other Adverse Events (participants affected / at risk) | 22/27 | 19/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Propranolol (N=27) | Placebo (N=27)
Vaso-occlusive crisis resulting in hospitalization (Musculoskeletal and connective tissue disorders) | 4 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Propranolol (N=27) | Placebo (N=27)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Atrioventricular (AV) block (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Drop in Blood Pressure (Cardiac disorders) | 0 | 1
Bilateral conjunctivitis (Eye disorders) | 0 | 1
Abdominal Paiin (Gastrointestinal disorders) | 1 | 2
Abdominal cramping (Gastrointestinal disorders) | 1 | 0
Abdominal pain and bloating (Gastrointestinal disorders) | 1 | 0
Blood per rectum (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2
Diarrhea, intermittent (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Nausea and vomiting (Gastrointestinal disorders) | 1 | 2
Stomach ache (Gastrointestinal disorders) | 1 | 1
Extreme tiredness (General disorders) | 0 | 2
Fatigue (General disorders) | 4 | 4
Feeling of internal heat (General disorders) | 1 | 0
Increased Fatigue (General disorders) | 1 | 0
Shakes (General disorders) | 0 | 1
E Coli Bacteremia (Infections and infestations) | 0 | 1
Fever (Infections and infestations) | 1 | 0
MRSA Positive (Infections and infestations) | 1 | 0
Sinus Infection (Infections and infestations) | 1 | 0
Sore throat (Infections and infestations) | 0 | 2
Sensitivity to cold (Metabolism and nutrition disorders) | 0 | 1
Pain Crisis (Musculoskeletal and connective tissue disorders) | 6 | 4
Pain, Back (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain, Bone (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain, Increased knee pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain, Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain, Joint (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain, Knee (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain, Left chest wall (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain, Leg (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain, Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain, back and chest (Musculoskeletal and connective tissue disorders) | 0 | 2
Toothache (Musculoskeletal and connective tissue disorders) | 0 | 1
Vaso-occlusive Crisis (Musculoskeletal and connective tissue disorders) | 2 | 2
Dizziness (Nervous system disorders) | 1 | 5
Headache (Nervous system disorders) | 8 | 8
Headache, extreme (Nervous system disorders) | 0 | 1
Worsening depression (Psychiatric disorders) | 0 | 1
Pylonephritis due to E. Coli (Renal and urinary disorders) | 0 | 1
Smelly urine and bladder spasms (Renal and urinary disorders) | 0 | 1
Delayed menstrual period (Reproductive system and breast disorders) | 0 | 1
Prolonged menstrual period (Reproductive system and breast disorders) | 0 | 1
Congestion, Upper Chest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Coughing, congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Sneezing/Allergies (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin abrasions due to pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Thrush (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atypical mycoplasma pneumonia, Suspected (Infections and infestations) | 1 | 0
Fracture, left foot (Musculoskeletal and connective tissue disorders) | 1 | 0
Fatigue with chest tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain, Hip (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain, Migrating (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain episode (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain, Right foot, plantar (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain, Leg, sharp shooting (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain, Shoulder/Chest (Musculoskeletal and connective tissue disorders) | 1 | 0
Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness/Vertigo (Nervous system disorders) | 1 | 0
Headache, Intermittent (Nervous system disorders) | 1 | 0
Lightheadness (Nervous system disorders) | 1 | 0
Vertigo (Nervous system disorders) | 1 | 0
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Shortness of breath on exertion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat, intermittent (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
sinus allergies (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Congestion, Sinus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat, worsening (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin abrasions due to pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
ED Visit (General disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes